CLINICAL TRIAL: NCT01560676
Title: A School-based Internet Obesity Prevention Program for Adolescents
Brief Title: Reducing Obesity and Type 2 Diabetes in High Risk Youth
Acronym: HEALTH[e]TEEN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Robin Whittemore, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1008007228
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Internet; School based; Obesity Prevention Program; Adolescents
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — galactosylceramide sulfotransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEALTH[e]TEEN (Active Comparator): 8 lessons over 6-8 weeks Education on healthy eating and physical activity Behavioral support for self-monitoring and goal setting
  Interventions: Behavioral: HEALTH[e]TEEN
- HEALTH[e]TEEN + CST (Active Comparator): 12 lessons over 6-8 weeks Education on healthy eating and coping skills training Behavioral support for self-monitoring and goal setting
  Interventions: Behavioral: HEALTH[e]TEEN + CST

INTERVENTIONS:
Behavioral: HEALTH[e]TEEN — 8 lessons over 6-8 weeks
  Arms: HEALTH[e]TEEN
Behavioral: HEALTH[e]TEEN + CST — 12 lessons over 6-8 weeks
  Arms: HEALTH[e]TEEN + CST

SUMMARY:
Compare the effect of the HEALT[e]TEEN program and a HEALTH[e]TEEN plus coping skills training delivered to high school students on BMI, nutrition and physical activity behaviors, and self-efficacy over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled in Health, Biology, or Public Health course

Exclusion Criteria:

* Cognitive ability unable to read or respond to questions in program

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 384 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
BMI | 6 months

SECONDARY OUTCOMES:
Dietary behavior | 6 months
  Healthy eating
Sedentary behavior | 6 months
  Computer, TV, video games
Physical activity | 6 months
  Moderate to vigorous exercise

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whittemore, PhD, Principal Investigator — Yale University; Margaret Grey, DrPH, Principal Investigator — Yale University
Locations (1):
- Yale, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Whittemore R, Jeon S, Grey M. An internet obesity prevention program for adolescents. J Adolesc Health. 2013 Apr;52(4):439-47. doi: 10.1016/j.jadohealth.2012.07.014. Epub 2012 Sep 27. PMID 23299003